CLINICAL TRIAL: NCT02766049
Title: Phase I/II Study of Anti-HIV Cellular Therapy Based on Dendritic Cells Pulsed With Chemically Inactivated Virus
Brief Title: Study of Anti-HIV Cellular Therapy Based on Dendritic Cells Pulsed With Chemically Inactivated Virus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAPPesq-0239/09
Record Dates: First submitted 2016-04-01; First posted 2016-05-09 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-05

CONDITIONS: HIV Infection
Keywords: HIV; immunotherapy; clinical trial; dendritic cell
MeSH Terms: conditions — HIV Infections

ARMS (3):
- (a) DC (Active Comparator): Autologous dendritic cells (3x10e7)
  Interventions: Biological: DC
- (b) DC 10e6+HIV-AT2 (Active Comparator): Autologous dendritic cells (3x10e6), pulsed with chemically inactive autologous HIV
  Interventions: Biological: DC10e6+HIV-AT2
- (c) DC 10e7+HIV-AT2 (Active Comparator): Autologous dendritic cells (3x10e7), pulsed with chemically inactive autologous HIV
  Interventions: Biological: DC10e7+HIV-AT2

INTERVENTIONS:
Biological: DC — Autologous dendritic cells (3x10e7)
  Arms: (a) DC
Biological: DC10e6+HIV-AT2 — Autologous dendritic cells (3x10e6), pulsed with chemically inactive autologous HIV
  Arms: (b) DC 10e6+HIV-AT2
Biological: DC10e7+HIV-AT2 — Autologous dendritic cells (3x10e7), pulsed with chemically inactive autologous HIV
  Arms: (c) DC 10e7+HIV-AT2

SUMMARY:
The aim of this study was to assess tolerability and safety of three different formulations of an anti-HIV immunotherapy based on autologous dendritic cells (DCs) pulsed with HIV chemically inactivated with Aldrithiol™-2 (AT-2). Patients were chronically infected with HIV, naïve for antiretroviral drugs. A possible immunological and virological favorable impact was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* patients with HIV infection;
* absence of antiretroviral therapy, antineoplastic therapy or the use of corticosteroids for at least six months prior to study entry;
* plasma viral load ≥ 1,000 copies / mL, stable (ie no variation > 0.5 log) in the six months before the start of the study;
* blood CD4+ T cells ≥ 350 /mL, stable (ie no variation > 25%) in the six months before the start of the study.

Exclusion Criteria:

* individuals without proper venous access for blood and apheresis collection procedure.
* use of drugs, alcohol, psychiatric disorder or any condition that interferes with the ability of patients to follow the requirements of the study;
* history of diagnosis of HIV infection <01 years;
* pregnancy or breast-feeding;
* use of antiviral therapy, in anticancer therapies or corticosteroids six months prior to study start;
* presence of chronic diseases, such as infection with hepatitis B (HBV) and C (HCV), human T-lymphotropic virus (HTLV) I / II or any condition that promotes immune system dysfunction, with the exception of HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with ≥ grade 3 adverse events related to product | 51 weeks
  AE graded by Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, version 1.0, December 2004

SECONDARY OUTCOMES:
Number of participants with change in plasma viral load from baseline, over the observation period | Baseline to 51 weeks
  Log10 change in HIV RNA
Number of participants with change in CD4+T cells from baseline, over the observation period | Baseline to 51 weeks
  Absolute number change of CD4+T cells

CONTACTS AND LOCATIONS:
Overall Officials: Alberto JS Duarte, Professor, Principal Investigator — University of Sao Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lu W, Arraes LC, Ferreira WT, Andrieu JM. Therapeutic dendritic-cell vaccine for chronic HIV-1 infection. Nat Med. 2004 Dec;10(12):1359-65. doi: 10.1038/nm1147. Epub 2004 Nov 28. PMID 15568033
- [Background] Oshiro TM, de Almeida A, da Silva Duarte AJ. Dendritic cell immunotherapy for HIV infection: from theory to reality. Immunotherapy. 2009 Nov;1(6):1039-51. doi: 10.2217/imt.09.68. PMID 20635918